CLINICAL TRIAL: NCT00448539
Title: An Open-Label Extension Study of Rufinamide Given as Adjunctive Therapy in Patients With Refractory Partial Seizures
Brief Title: Open-Label Extension Study of Rufinamide Given as Adjunctive Therapy in Patients With Refractory Partial Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early by the sponsor due to the discontinuation of clinical development for rufinamide.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2080-A001-302; 2016-004950-14 (EudraCT Number)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Refractory Partial Onset Seizures
Keywords: Refractory Partial Onset Seizures, epilepsy
MeSH Terms: conditions — Epilepsy | interventions — rufinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rufinamide (Rufinamide During Core Study) (Experimental)
  Interventions: Drug: Rufinamide
- Rufinamide (Placebo During Core Study) (Experimental)
  Interventions: Drug: Rufinamide

INTERVENTIONS:
Drug: Rufinamide — Dose will be maintained within the range of 2400 to 4800 mg/day (i.e., 1200 to 2400 mg twice daily).
  Other Names: E2080

SUMMARY:
This was an open-label extension study in adolescent and adult (between 12 and 80 years old) participants who had completed their participation in Study E2080-A001-301. The main objective of this study was to evaluate the safety and efficacy of long-term administration of rufinamide for the control of epileptic seizures in participants who had refractory partial seizures despite treatment with a maximum of three approved antiepileptic drugs (AEDs).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Completion of Study E2080-A001-301 and full compliance with the inclusion and exclusion criteria for that study (excluding criteria that are related to seizure occurrences).
2. Patient willing to participate and written consent signed by patient or legal guardian provided prior to entering this study or undergoing any study procedures. In addition, if the patient is unable to provide written informed consent and it is provided by a legal guardian, assent of the patient (if the patient is able) must also be obtained.
3. Female patients of non-childbearing potential by reason of surgery, radiation, or menopause (at least one year post onset); female patients of childbearing potential who are using at least two approved methods of contraception (such as an intrauterine device [IUD], implant, oral contraceptive, or barrier method plus spermicide). Use of a low-dose estrogen oral contraceptive alone will not be permitted. Female patients of childbearing potential must agree to continue to use two approved methods of contraception through the follow-up visit or for 30 days after their final dose of study medication, whichever is longer.

EXCLUSION CRITERIA:

1. Discontinuation from Study E2080-A001-301 for any reason, before the termination of the study.
2. Evidence of non-compliance with study drug or ongoing AED dosing during Study E2080-A001-301.
3. Evidence of clinically significant disease (cardiac, respiratory, gastrointestinal, hepatic (e.g., ALT > 3x ULN), hematologic, renal, or psychiatric disease, etc.) that in the opinion of the Investigator could affect the patient's safety or trial conduct.
4. Progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
5. History of alcohol abuse in the past 2 years.
6. History of suicide attempt within the previous 10 years.
7. Multiple drug allergies (dematological, heatological or organ toxicity) or more than one severe drug reaction.
8. Concomitant use of felbamate or vigabatrin.
9. Pregnancy.
10. Clinically significant ECG abnormality.
11. All patients with a diagnosis of Congenital Short QT Syndrome. Patients with a family history of Congenital Short QT Syndrome may be excluded on the basis of the Investigator's clinical judgement.
12. Presence of major active psychiatric disorder. Patients will be allowed who are taking a stable dose of selective serotonin reuptake inhibitor (SSRI) or mixed serotonin and norepinephrine uptake inhibitor antidepressant.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2007-03-15 (Actual); Primary Completion 2010-05-14 (Actual); Study Completion 2010-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Bradenton Research Center, Bradenton, Florida
  - University of Florida, The Neuroscience Institute at Shands, Jacksonville, Florida
  - Pediatric Neurologists of Palm Beach, Loxahatchee Groves, Florida
  - Pediatric Neurosciences, PA, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Child Neurology Associates, PC, Atlanta, Georgia
  - Southern Illinois University Neurology and Pharmacology, Springfield, Illinois
  - McFarland Clinic PC, Ames, Iowa
  - John Hopkins Hospital, Dept. of Neurology, Baltimore, Maryland
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Dartmouth Medical School Neuroscience Center, Lebanon, New Hampshire
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - New York University Medical Centre, Comprehensive Epilepsy Center, New York, New York
  - Weill Cornell Medical Center, Comprehensive Epilepsy Center, New York, New York
  - Asheville Neurology Specialists, Asheville, North Carolina
  - Ohio State University, Columbus, Ohio
  - Medical University of Ohio at Toledo - Dept. of Neurology, Toledo, Ohio
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania Medical Center-Department of Neurology, Philadelphia, Pennsylvania
  - University of Tennessee Health Sciences Center, Dept. of Neurology, Memphis, Tennessee
  - Access Clinical Trials, Inc, Nashville, Tennessee
  - Neurological Clinic of Texas, P.A., Dallas, Texas
  - Texas Tech University Health Sciences Center, Dept. of Neuropsychiatry, El Paso, Texas
  - Fletcher Allen Healthcare, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed double-blind study E2080-A001-301 were allowed to enter in open-label extension Study 302. Participants completed a 12-day Transition Phase in Study 301 and received the same rufinamide maintenance dose that they achieved in Study 301 (Arm1), or transitioned from placebo to 3200 mg/day, beginning at 800 mg/day (Arm2).
Pre-assignment Details: Four participants who intended to enroll from Study 301 to 302 did not enroll and were considered screening failures.
Groups:
- Rufinamide (Rufinamide During Core Study): Participants entered this open-label extension study from E2080-A001-301 double-blind core study, where they received rufinamide in the core study. Prior to starting the extension study, participants completed a 12-day Transition Phase. For participants who immediately entered study 302 after study 301, rufinamide was maintained at dose of 2400 or 3200 milligram per day (mg/day) achieved at the end of study 301. Participants with delay between the end of Study 301 and the beginning of Study 302 started rufinamide at a dose of 800 mg/day, and had the dose titrated to the maximum tolerated dose (2400 or 3200 mg/day) over the next 12 to 18 days. During the open-ended open-label Maintenance Phase, changes in the rufinamide dose were permitted for all participants; however, the dose was maintained within the range of 2400 to 4800 mg/day (i.e., 1200 to 2400 mg twice daily).
- Rufinamide (Placebo During Core Study): Participants entered this open-label extension study from E2080-A001-301 double-blind core study, where they received placebo in the core study. Prior to starting the extension study, participants completed a 12-day Transition Phase where they transitioned from placebo to rufinamide at 800 mg/day at the start of transition phase, with subsequent dose increased to 3200 mg/day. During the open-ended open-label Maintenance Phase, changes in the rufinamide dose were permitted for all participants; however, the dose was maintained within the range of 2400 to 4800 mg/day (i.e., 1200 to 2400 mg twice daily).
Period: Overall Study
Arm/Group | Rufinamide (Rufinamide During Core Study) | Rufinamide (Placebo During Core Study)
Started | 134 | 152
Completed | 0 | 0
Not Completed | 134 | 152
Not completed — Medication non-compliance | 4 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Request of the investigator or sponsor | 67 | 54
Not completed — Withdrawal by Subject | 20 | 24
Not completed — Diary non-compliance | 1 | 0
Not completed — Adverse Event | 9 | 26
Not completed — Lack of Efficacy | 27 | 40
Not completed — Miscellaneous | 2 | 1
Not completed — Change of meds | 2 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Rufinamide (Rufinamide During Core Study): Participants entered this open-label extension study from E2080-A001-301 double-blind core study, where they received rufinamide in the core study. Prior to starting the extension study, participants completed a 12-day Transition Phase. For participants who immediately entered study 302 after study 301, rufinamide was maintained at dose of 2400 or 3200 mg/day achieved at the end of study 301. Participants with delay between the end of Study 301 and the beginning of Study 302 started rufinamide at a dose of 800 mg/day, and had the dose titrated to the maximum tolerated dose (2400 or 3200 mg/day) over the next 12 to 18 days. During the open-ended open-label Maintenance Phase, changes in the rufinamide dose were permitted for all participants; however, the dose was maintained within the range of 2400 to 4800 mg/day (i.e., 1200 to 2400 mg twice daily).
- Total: Total of all reporting groups
Arm/Group | Rufinamide (Rufinamide During Core Study) | Rufinamide (Placebo During Core Study) | Total
Number analyzed (Participants) | 134 | 152 | 286
Age, Customized [Number; unit: participants] — Safety population
  participants
    12 to <18 years | 6 | 18 | 24
    18 to <65 years | 123 | 129 | 252
    >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population: All participants who received at least 1 dose of study medication.
  Participants
    Female | 63 | 80 | 143
    Male | 71 | 72 | 143
Race/Ethnicity, Customized [Number; unit: participants] — Race (safety population)
  participants
    Black | 7 | 13 | 20
    White | 115 | 121 | 236
    Hispanic | 10 | 11 | 21
    Native American | 0 | 2 | 2
    Asian/Pacific Islander | 2 | 2 | 4
    Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Total Partial Seizure Frequency Per 28 Days Relative to the Baseline Phase
Description: Seizure data was collected via patient diaries. "OL" refers to "open-label."
Time Frame: Baseline, Titration Phase (Days 1 to 18), Maintenance Phase
Population: Intent-to-treat (ITT) population: All subjects who completed titration to open-label medication
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Rufinamide (Rufinamide During Core Study) | Rufinamide (Placebo During Core Study)
Number analyzed (Participants) | 134 | 151
Percentage change
  OL Titration Phase | -35.65 [-100.0 to 1570.7] | -45.10 [-100 to 518.2]
  OL Maintenance Phase | -30.95 [-100.0 to 246.5] | -31.10 [-100 to 322.4]

ADVERSE EVENTS:
Time Frame: From the date of first dose of rufinamide through study termination (up to 3 years and 10 months)
Arm/Group | Rufinamide (Rufinamide During Core Study) | Rufinamide (Placebo During Core Study)
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/152
Serious Adverse Events (participants affected / at risk) | 29/134 | 23/152
Other Adverse Events (participants affected / at risk) | 88/134 | 114/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (Rufinamide During Core Study) (N=134) | Rufinamide (Placebo During Core Study) (N=152)
Myocardial infarction (Cardiac disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 2
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Ventriculoperitoneal shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 5 | 7
Dysarthria (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Grand Mal Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0
Postictal state (Nervous system disorders) | 0 | 2
Status epilepticus (Nervous system disorders) | 3 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Epileptic psychosis (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (Rufinamide During Core Study) (N=134) | Rufinamide (Placebo During Core Study) (N=152)
Diplopia (Eye disorders) | 4 | 10
Abdominal pain upper (Gastrointestinal disorders) | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 12 | 19
Vomiting (Gastrointestinal disorders) | 14 | 12
Fatigue (General disorders) | 6 | 15
Pyrexia (General disorders) | 1 | 9
Sinusitis (Infections and infestations) | 12 | 8
Upper respiratory tract infection (Infections and infestations) | 9 | 6
Contusion (Injury, poisoning and procedural complications) | 8 | 4
Fall (Injury, poisoning and procedural complications) | 7 | 5
Skin laceration (Injury, poisoning and procedural complications) | 9 | 5
Weight decreased (Metabolism and nutrition disorders) | 8 | 9
Decreased appetite (Metabolism and nutrition disorders) | 2 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Convulsion (Nervous system disorders) | 10 | 20
Dizziness (Nervous system disorders) | 11 | 43
Headache (Nervous system disorders) | 15 | 17
Somnolence (Nervous system disorders) | 2 | 14
Anxiety (Psychiatric disorders) | 7 | 6
Depression (Psychiatric disorders) | 12 | 3
Insomnia (Psychiatric disorders) | 13 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Coordination Abnormal (Nervous system disorders) | 4 | 10

LIMITATIONS AND CAVEATS:
This study was terminated early by the sponsor due to the discontinuation of clinical development for rufinamide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No